CLINICAL TRIAL: NCT05423613
Title: Randomized Controlled Evaluator-blinded Trial of Microneedling for the Treatment of Hypertrophic Scars of Adult Burn Survivors and Patients With Severe Skin Disorders
Brief Title: Microneedling for Burn Hypertrophic Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Bernadette Nedelec, Full professor, McGill University, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20.184
Record Dates: First submitted 2022-06-02; First posted 2022-06-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Burn Scar
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microneedling treated scar (Experimental): Microneedling
  Interventions: Procedure: Microneedling
- Control scar (No Intervention): No intervention, standard of care

INTERVENTIONS:
Procedure: Microneedling — A 5% lidocaine anesthetic cream will be applied to the scar to be treated and will be wrapped with an occlusive dressing (saran wrap) for 30 minutes prior to the procedure. The same scar will be subjected to the ACS-Pen treatment at a depth of 1.5 mm or less depending on the results of the thickness measurement performed prior to treatment. Within 5 minutes after the microneedling treatment, a thin layer of triamcinolone acetonide and 2% xylocaine (1:3 ratio) suspension will be spread over the scar. The physician will then gently massage the product into the microneedling columns. The same amount will be used for each subsequent treatment. The patient will also be given a small amount of hydrocortisone 2.5% (low potency corticosteroid) to be applied to the treated site at 12 hours and 24 hours post-treatment.
  Arms: Microneedling treated scar

SUMMARY:
Approximately 33 to 91% of severe burn victims will develop hypertrophic scars. Hypertrophic scars are defined as erythematous (red), raised and rigid scars that can cause pain and itching, among other things. They cause psychological distress and affect the quality of life of burn victims. Microneedling is a technique that uses an electrical device to create hundreds of microchannels that penetrate the skin layers. This study is interested in determining the effectiveness of microneedling in improving the pliability, thickness and erythema of hypertrophic scars. Each scar will receive up to 5 ACS-pen treatments followed by the application of cortisone (triamcinolone acetonide). Knowing that microneedling increases the absorption of products applied to the skin by about 80%, it is logical to think that creating these channels to the dermis and applying cortisone afterwards would have a beneficial effect on the hypertrophic scars of these patients.

DETAILED DESCRIPTION:
Patients will receive microneedling once every six weeks for a maximum of five treatments

ELIGIBILITY:
Inclusion Criteria:

* Any gender or race
* 16 years of age or older
* Have at least 2 HSc that meet the clinical criteria for HSc
* Provide written informed consent.

Exclusion Criteria:

* Patients with keloid scars
* Mature scar site
* A psychiatric condition or cognitive impairment that interferes with their ability to follow the treatment protocol
* Dermatological conditions (i.e. psoriasis, eczema, etc.) in the area of the evaluation site
* An allergy to ultrasound gel
* On anticoagulant medications
* Inability to understand English or French.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Skin Erythema Changes | Baseline, before treatments #3, #4 and #5, post 6 weeks and 12 weeks
  Erythema index measure by Mexameter, values from 0 to 999. The erythema values are individual for each person and depend strongly on the ethnic group. The measurements are generally used to determine changes before and after a treatment.
Cutometer Skin Elasticity Changes | Baseline, before treatments #3, #4 and #5, post 6 weeks and 12 weeks
  Skin elasticity measures (r0- Cutometer), mm
Skin Thickness Changes | Baseline, before treatments #3, #4 and #5, post 6 weeks and 12 weeks
  Ultrasound skin measures, mm

SECONDARY OUTCOMES:
Patient reported effectiveness of intervention | Baseline, 12 weeks post intervention
  Visual analog scale (score 0-none to 10-worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Villa Medica Rehabilitation Hospital, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No